CLINICAL TRIAL: NCT04227834
Title: Re-infection Rates of Soil-transmitted Helminth Infections Among School-aged Children Following a Single or a 4-monthly Health Hygiene Education: an Open Label Clinical Trial
Brief Title: Soil-transmitted Helminth Reinfection Rates After Single and Repeated School Hygiene Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Inke Nadia Diniyanti Lubis, Head of Tropical Medicine Master Programme, Universitas Sumatera Utara
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STH032019
Record Dates: First submitted 2020-01-04; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Helminthiasis; Ascaris Infection; Trichuris Infection; Hookworm Infections; Children, Only
Keywords: Soil-transmitted helminth; School-aged children; Health hygiene; Education
MeSH Terms: conditions — Helminthiasis; Ascariasis; Trichuriasis; Hookworm Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single education (Active Comparator): Single health hygiene education
  Interventions: Behavioral: Health hygiene education
- Repeated education (Experimental): Four-monthly health hygiene education
  Interventions: Behavioral: Health hygiene education

INTERVENTIONS:
Behavioral: Health hygiene education — A cartoon video explaining the etiology, risk factors, clinical symptoms, treatment and prevention of helminthiasis were given to the school-aged children

SUMMARY:
Soil-transmitted helminth (STH) infections caused by Ascaris lumbricoides, Trichuris trichiura, or hookworm, affect approximately 1.5 millions individuals primarily in tropical and subtropical regions. STHs infections have been associated with delay in growth and development in children. The prevalence in Indonesia varied from 45% to 65%, but in poor sanitation areas the prevalence can increased to 80%. World Health Organization currently recommends mass treatment with benzimidazoles and health hygiene education to control the disease. In this study we evaluated the effectiveness of single and four-monthly health hygiene education to STH reinfection rates among school-aged children in Mandailing Natal district, North Sumatera province, Indonesia.

DETAILED DESCRIPTION:
In this study we evaluate the prevalence of STH among school-aged children using Kato Katz examination prior to enrolment to the study. Two elementary schools in Mandailing Natal district, North Sumatera province, Indonesia have been selected and received either a single or repeated health hygiene education. Preliminary knowledge was also assessed using a questionnaire. Infected children received treatment of albendazole 400 mg for 3 days. Evaluation on reinfection status and STH knowledge is done at 4 month, 8 month and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children who are negative for STHs infection on Kato Katz examination following 3 days treatment of albendazole

Exclusion Criteria:

* Parents who refused to participate in the study
* Severe malnutrition
* Co-infected with other helminth infections

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 432 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2020-03-02 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of repeated health hygiene education on the reinfection rates of STHs among school-aged children | 12 months
  STH prevalence at 12 months

SECONDARY OUTCOMES:
Prevalence of STHs among school-aged children prior to intervention | STH prevalence at month 0
  Ascaris lumbricoides, Trichuris trichiura, hookworm infections at month 0
Knowledge of STHs prevention measures among school-aged children before and after intervention | 12 months
  A questionnaire used to evaluate the knowledge about STHs prevention

CONTACTS AND LOCATIONS:
Overall Officials: Rizky KA Nasution, MD, Principal Investigator — Universitas Sumatera Utara
Locations (1):
- Singkuang sub-district, Mandailing Natal district, Panyabungan, North Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT04227834/Prot_000.pdf
  • Informed Consent Form (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT04227834/ICF_001.pdf